CLINICAL TRIAL: NCT01663883
Title: Optic Nerve Head Autoregulation During Changes in Arterial Blood Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Gerhard Garhofer, Ass. Prof. Priv. Doz. Dr., Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: OPHT-210911
Record Dates: First submitted 2012-01-24; First posted 2012-08-13 (Estimated); Last update posted 2012-08-13 (Estimated); Status verified 2012-08

CONDITIONS: Decreased Vascular Flow
Keywords: Blood flow autoregulation; optic nerve head blood flow; isometric exercise; Autoregulation; ocular physiology
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Healthy subjects (Experimental)
  Interventions: Other: Isometric exercise

INTERVENTIONS:
Other: Isometric exercise — use of a handgrip for 3x2 minutes

SUMMARY:
Constant despite changes in perfusion pressure. It is observed in many vascular beds of the human body to prevent that variations in perfusion pressure are directly transmitted into changes in blood flow. This is necessary to prevent ischemia and/or hypoxia during decreased blood flow and bleeding or increased capillary pressure during increased blood flow.

In the eye, several studies have reported that retinal blood flow is autoregulated over a wide range of ocular perfusion pressures. Unfortunately only few data are available for the optic nerve head. To gain data about autoregulation is of special importance given that several important ocular diseases such as glaucoma and age-related macular degeneration are associated with impaired autoregulation. In humans most data were collected using laser Doppler flowmetry.

The present study aims to investigate the phenomenon of transient reduction in blood flow and to gain insight in the regulatory mechanisms of optic nerve head blood flow during isometric exercise.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged between 18 and 35 years, nonsmokers
* Normal findings in the medical history and physical examination unless the investigator considers an abnormality to be clinically irrelevant
* Normal ophthalmic findings, ametropia less than 3 diopters

Exclusion Criteria:

* Regular use of medication, abuse of alcoholic beverages, participation in a clinical trial in the 3 weeks preceding the study
* Treatment in the previous 3 weeks with any drug (except oral contraceptives)
* Symptoms of a clinically relevant illness in the 3 weeks before the first study day
* Blood donation during the previous 3 weeks

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2012-02; Primary Completion 2012-04 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Optic nerve head blood flow | 12 minutes

SECONDARY OUTCOMES:
Systolic/diastolic blood pressure | 14 minutes
Intraocular pressure | at baseline and minute 13
Pulse rate | 14 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Garhöfer, MD, Principal Investigator — Department of Clinical Pharmacology, Medical University of Vienna
Locations (1):
- Department of Clinical Pharmacology, Vienna, Vienna, Austria